CLINICAL TRIAL: NCT02072967
Title: Observational Program for Evaluation of Ribomustin and Rituximab Combined Therapy With Following Rituximab Maintenance of Relapsed or Refractory Indolent B-cell Non-Hodgkin's Lymphoma
Brief Title: Ribomustin in the Second Line Therapy of Relapsed or Refractory Indolent B-cell Non-Hodgkin's Lymphoma
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: RU-BEN-NI-001
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Relapsed; Refractory; Non-Hodgkin Lymphoma; Bendamustine
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence | interventions — Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ribomustin and rituximab
  Interventions: Other: Ribomustin; Other: rituximab

INTERVENTIONS:
Other: Ribomustin — Routine practice
  Other Names: bendamustine
Other: rituximab — Routine practice
  Other Names: Mabthera

SUMMARY:
Prospective multicenter observational non-interventional study to assess routine clinical practice of Bendamustine use in the second line therapy of relapsed or refractory indolent B-cell non-Hodgkin's lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Doctor's decision to prescribe Ribomustin and rituximab combined therapy for the treatment of relapsed or refractory indolent B-cell Non-Hodgkin's Lymphoma (iNHL)
* Informed Consent Form for personal data handling signed by the program participant, authorized by the Independent Ethics Committee
* Eastern Cooperative Oncology Group (ECOG) status < 2.
* Confirmed relapse or disease progression of B-cell CD20+ Non-Hodgkin's Lymphoma (lymphocytic, lymphocytoplasmocytic, follicular, marginal zone) after minimum one line of iNHL treatment
* Patients with relapsed or refractory indolent B-cell Non-Hodgkin's Lymphoma with current or planned Ribomustin and rituximab combined therapy with following rituximab maintenance therapy

Exclusion Criteria:

* Indolent Non-Hodgkin's Lymphoma transformation
* Lymphoma with central nervous system (CNS) involvement
* Presence of second malignant tumor.
* Currently participating in any clinical trial, and/or has taken an investigational drug within 28 days prior to enrollment.
* Contraindications for Ribomustin usage in accordance with product label
* Contradictions for rituximab usage in accordance with product label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Relapsed or Refractory Indolent B-cell Non-Hodgkin's Lymphoma with planned combined Ribomustin and rituximab therapy
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2012-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 90 days post-treatment

SECONDARY OUTCOMES:
Adverse drug reactions | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (35):
- Russia (35):
  - City Clinical Hospital #8, Barnaul
  - Chelyabinsk Regional Oncology Dispensary/15, Chelyabinsk
  - Vologda Regional Clinical Hospital #2, Cherepovets
  - Regional Oncology Dispensary/35, Irkutsk
  - Irkutsk Regional Сlinical Hospital/31, Irkutsk
  - Kaluga Regional Clinical Hospital/02, Kaluga
  - District Cancer center od Khanty -Mansiysk, Khanty-Mansiysk
  - City Сlinical Hospital#7/25, Krasnoyarsk
  - Regional Сlinical Hospital/12, Krasnoyarsk
  - Adygei Regional Clinical Oncology Dispensary/11, Maykop
  - Scientific Medical Surgical Center n.a.I.V.Pyrogov/17, Moscow
  - European Medical Center, Moscow
  - RONC n.a.N.N.Blokhin/18, Moscow
  - Сentral Clinical Hospital n.a. Semashko N.A./30, Moscow
  - Moscow Scientific Research Oncology Institution n.a.P.A. Gertzen/37, Moscow
  - Central Clinical Hospital of Department of Presidential Affairs, Moscow
  - Municipal Сlinical Hospital № 12/20, Nizhny Novgorod
  - Novosibirsk State Regional Clinical Hospital/23, Novosibirsk
  - Medical Radiology Scientific Center/38, Obninsk
  - Omsk Regional Clinical Hospital/40, Omsk
  - City Сlinical Hospital#1 n.a.Kabanov A.N./13, Omsk
  - Orenburg State Medical Academy/05, Orenburg
  - Rostov Scientific Research Oncology Institution/01, Rostov-on-Don
  - City Сlinical Oncological Dispensary/22, Saint Petersburg
  - City Сlinical Hospital#31/08, Saint Petersburg
  - Military-Medical Academy n.a. Kirova, Saint Petersburg
  - Scientific Research Oncological Institution n.a. Petrov N.N./29, Saint Petersburg
  - Samara State Medical University' Clinics/36, Samara
  - Road Clinical Hospital on Rostov-Main Station OAO RZhD/06, Smolensk
  - Surgut Regional Clinical Hospital, Surgut
  - Tula Regional Clinical Hospital/21, Tula
  - Volgograd Regional Clinical Oncology Dispensary#1/10, Volgograd
  - Vologda Regional Clinical Hospital/39, Vologda
  - Yekaterinburg Regional Clinical Hospital #1, Yekaterinburg
  - Sakhalin Regional Oncology Dispensary/32, Yuzhno-Sakhalinsk

IPD SHARING:
Plan to Share IPD: Undecided